CLINICAL TRIAL: NCT03038126
Title: Care Coordination/Telehealth to Address Patient Safety and Poor Outcomes in CKD
Brief Title: Care Coordination/Home Telehealth to Safeguard Care in CKD
Acronym: CCHT in CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Baltimore VA Medical Center (U.S. Federal Agency); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jeffrey Fink, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HP-00058634; R34DK102177 (NIH)
Record Dates: First submitted 2017-01-29; First posted 2017-01-31 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Safety Issues; Chronic Kidney Disease
Keywords: chronic kidney disease; patient safety; home telehealth
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CCHT (Active Comparator): Veterans Administration (VA) CCHT with an established guideline-based CKD DMP, augmented laboratory monitoring, and decision support from the VA Renal Inter-disciplinary Safety clinic (RISC).
  Interventions: Other: CCHT
- Usual care (Placebo Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: CCHT — Veterans Administration (VA) CCHT program available to veterans with difficult to manage chronic conditions and employing an established guideline-based CKD DMP, augmented laboratory monitoring, and decision support from the VA Renal Inter-disciplinary Safety clinic (RISC).
  Arms: CCHT
Other: Usual care — Standard clinical care
  Arms: Usual care

SUMMARY:
Home telehealth monitoring of veterans with chronic kidney disease, with a disease management protocol and safety-specific decision support, will increase the detection of adverse safety events, and in turn, reduce the need for urgent health resource utilization and associated poor outcomes.

DETAILED DESCRIPTION:
Pre-dialysis chronic kidney disease (CKD) is associated with a high risk of harm related to medical care (adverse safety events). These events may occur outside the purview of the medical system, and hence, are under-recognized. Health information technology (IT) can enhance the detection of such events, and coordinated care can prevent their adverse consequences. Study design: 6-month randomized trial of coordinated care/home telehealth (CCHT) vs usual care in CKD patients. Intervention: Veterans Administration (VA) CCHT with a guideline-based CKD DMP, augmented laboratory monitoring, and decision support from the VA Renal Inter-disciplinary Safety clinic (RISC). Study population: Veterans with Stage III-V CKD (no expected dialysis within 6 months), age ≥ 60 years old, and diabetes (n = 65 per arm). Study Site: Baltimore VA Medical Center (BVAMC), VA Geriatrics Research, Education and Clinical Center (GRECC), and RISC. Specific Aim 1: Compare detection of adverse safety events in CKD patients assigned to CCHT vs usual care. Specific Aim 2: Compare the frequency of urgent health service use and participant satisfaction with CCHT vs usual care group. Study Measurements: Vital sign and clinical measurements (daily BP, weight, and finger stick glucose), laboratory values, and patient- reported safety events obtained per CCHT protocol vs patient-reported safety events, laboratory values, and assessment at a mid-study safety clinic visit in usual care protocol. Emergency department (ED) visits, hospitalization, renal progression, incidence of ESRD, and death will be measured in both groups along with patient satisfaction. Outcomes: Aim 1: Counts of a diverse set of adverse safety events including hypoglycemia, hypotension, volume loss (by weight change), hyperkalemia, acute kidney injury (AKI), and patient-reported safety incidents. Aim 2: ED visits, hospitalization, and other adverse outcomes including renal function loss, ESRD, and death. Analytic plans: Adjusted rates of events tracked in Aim 1 and 2 and expressed as counts per month will be compared in CCHT vs usual care group with multivariate models as indicated. Expected findings: CCHT will increase the detection of adverse safety events but reduce urgent health resource utilization and adverse outcomes. Public Health Relevance: Home telemonitoring of CKD patients in conjunction with coordinated care and decision support can increase the detection of adverse safety events that occur outside the traditional health care system and offer new opportunities to reduce their associated poor outcomes on a platform that allows ready dissemination across a national health network.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with Stage III-V CKD
* Diabetes

Exclusion Criteria:

* Expectation of dialysis or death within 6 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CCHT | Usual Care
Started | 63 | 55
Completed | 54 | 51
Not Completed | 9 | 4
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Long Term Hospitalization | 2 | 0
Not completed — Too Ill to Participate | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CCHT | Usual Care | Total
Number analyzed (Participants) | 63 | 55 | 118
Age, Continuous [Mean (Standard Deviation); unit: year] | 70.9 (5.4) | 70.7 (6.2) | 70.8 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 53 | 114
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 37 | 36 | 73
  White | 24 | 17 | 41
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 63 | 55 | 118
eGFR [Mean (Standard Deviation); unit: ml/min/1.73m2] | 42.5 (12.7) | 42.4 (13.9) | 42.5 (13.2)

OUTCOME MEASURES:

1. Primary Outcome: Safety Events
Description: number of safety events discovered in each study arm. In-center safety events include those detected during study visit vital signs and laboratory results (e.g. hypotension, hyperkalemia, etc.) Self-reported safety events include patient-identified incidents reported to staff at study visits (e.g. hypoglycemia, leg/ankle swelling, falls etc.)
Time Frame: 3 months, 6 months
Population: number analyzed in each row differs due to various reasons including inability to complete specific measurements, missed visits, drop-out, ESRD, death, and loss to follow-up.
Measure: Number; unit: safety events
Arm/Group | CCHT | Usual Care
Number analyzed (Participants) | 63 | 55
safety events
  Self-Reported Safety Events (3 months): number analyzed (Participants) | 55 | 52
  Self-Reported Safety Events (3 months) | 70 | 54
  Self-Reported Safety Events (6 months): number analyzed (Participants) | 54 | 53
  Self-Reported Safety Events (6 months) | 61 | 58
  In-Center Safety Events (3 months): number analyzed (Participants) | 53 | 48
  In-Center Safety Events (3 months) | 30 | 30
  In-Center Safety Events (6 months): number analyzed (Participants) | 51 | 48
  In-Center Safety Events (6 months) | 26 | 28

2. Secondary Outcome: Change in Renal Function
Description: Change in GFR from baseline to 6 months
Time Frame: 6 months
Population: number analyzed differs from total population due to various reasons including inability to complete specific measurements, missed visits, drop-out, ESRD, death, and loss to follow-up.
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Arm/Group | CCHT | Usual Care
Number analyzed (Participants) | 61 | 53
ml/min/1.73m2 | -0.36 (6.44) | -3.19 (9.44)

3. Secondary Outcome: Hospitalization
Description: Frequency of unanticipated hospitalization events over duration of study
Time Frame: 3 months, 6 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: hospitalizaztions per month
Arm/Group | CCHT | Usual Care
Number analyzed (Participants) | 63 | 55
hospitalizaztions per month
  Reported at 3 month visit: number analyzed (Participants) | 55 | 52
  Reported at 3 month visit | 0.11 [0.07 to 0.17] | 0.14 [0.08 to 0.27]
  Reported at 6 month visit: number analyzed (Participants) | 54 | 53
  Reported at 6 month visit | 0.11 [0.07 to 0.18] | 0.15 [0.10 to 0.23]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the duration of study participation up to 6 months per participant or censor if earlier
Arm/Group | CCHT | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/63 | 1/55
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/55
Other Adverse Events (participants affected / at risk) | 49/63 | 51/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CCHT (N=63) | Usual Care (N=55)
In-Center Hypoglycemia (Endocrine disorders) | 7 | 7 — Blood glucose < 70 with or without symptoms. Detected on study visit labs.
In-Center Hyperglycemia (Endocrine disorders) | 2 | 3 — Blood Glucose >350 mg/dL. Detected on study visit labs.
In-Center Hypotension (Cardiac disorders) | 11 | 10 — Systolic Blood Pressure < 90 mmHg or Diastolic Blood Pressure < 45 mmHg. Detected during study visit vital signs.
In-Center Orthostasis (Cardiac disorders) | 30 | 36 — Drop >20 mmHg from sitting blood pressure to standing blood pressure and/or increase >15 bpm from sitting pulse to standing pulse. Detected during study visit vital signs.
Patient-Reported Hyperkalemia (Renal and urinary disorders) | 5 | 4 — Patient-reported high potassium blood level that required a change in medication, change in diet, and/or taking a prescription of kayexelate or polystyrene.
Patient-Reported Dizziness (General disorders) | 5 | 7
Patient-Reported Falls (General disorders) | 3 | 4
Patient-Reported Bleeding (Blood and lymphatic system disorders) | 2 | 5
Patient-Reported Nausea, Vomiting, and/or Diarrhea (Gastrointestinal disorders) | 9 | 8
Patient-Reported New or Worseneing Ankle Swelling (Cardiac disorders) | 10 | 10
Patient-Reported Muscle Weakness or Cramps (General disorders) | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT03038126/SAP_000.pdf
  • Study Protocol (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT03038126/Prot_001.pdf